CLINICAL TRIAL: NCT05519748
Title: Effectiveness of an Online Psychoeducation Program for Improving Coping in People With a High Level of Dissociative Symptoms: A Pilot Randomized Waitlist-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Sigma Theta Tau International Honor Society of Nursing (Other)
Responsible Party: Principal Investigator, Lam Kam Ki Stanley, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6906334
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Dissociation
MeSH Terms: conditions — Dissociative Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online psychoeducational program (Experimental): The intervention group will receive an online psychoeducational program for 8 weeks. The psychoeducation package consists of 16 different sets of reading materials and post-session writing/reflection exercises, which will be delivered to the participants twice a week. The program is designed to be a brief, trauma-informed, dissociation-focused education package that aims to enable users to better understand and cope with their post-traumatic and dissociative reactions and related life challenges. There are specific psychoeducation elements in each session, such as: (1) safety issues planning, (2) understanding the impacts of trauma and stress, (3) understanding the concept of dissociation and integration of the personality, (4) identifying and coping with the post-traumatic and dissociative symptoms, (5) identifying trauma-related cognitive distortions.
  Interventions: Behavioral: Online psychoeducational program
- Waitlist control (Other): The waitlist control group will receive an online psychoeducational program for 8 weeks a week after the completion of the two-month follow-up in the intervention group. The psychoeducation package is identical to the program in the intervention group.
  Interventions: Behavioral: Online psychoeducational program

INTERVENTIONS:
Behavioral: Online psychoeducational program — The intervention group will receive an online psychoeducational program for 8 weeks. The psychoeducation package consists of 16 different sets of reading materials and post-session writing/reflection exercises, which will be delivered to the participants twice a week.

SUMMARY:
Subject Population Our study's target population is people with pathological dissociation in the community.

Research Design A pilot randomized waitlist-controlled trial will investigate the effects of an online psychoeducation program on coping, symptom management, and self-efficacy of people with pathological dissociation immediately (posttest-1) and 2-month (posttest-2) post-intervention. Supplementary semi-structured interviews will be conducted for process evaluation. The analysis and reporting of the trial will strictly follow the CONSORT guidelines.

Instrument The primary outcome of our study is the coping ability of individuals with pathological dissociation, which will be assessed by the Brief Coping Orientation to Problems Experienced Inventory (Brief-COPE). The secondary outcome measures are dissociative symptoms, emotional regulation, and self-efficacy, which would be assessed by the Dissociative Experiences Scale-Taxon (DES-T), the Emotion Regulation Questionnaire (ERQ), and the General Self-Efficacy Scale (GSES) accordingly.

Procedure The online psychoeducation program is developed based on an integrative theoretical framework that integrates the Stress and Coping model, Cognitive-Behavioural Theory, Bandura's self-efﬁcacy theory, and findings of our previous feasibility studies on this psychoeducational program. Participants will be recruited via posting on social media and online forums. A 16-session online psychoeducation program will be delivered to the participants in eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* agree to give informed consent and participate
* aged 18 or above
* self-reported symptoms or experiences of pathological dissociation
* screened positive on the Chinese version of the DES-T (i.e., DES-T score 20 or above) at a baseline screening
* able to understand and communicate in Chinese-Cantonese
* have access to the internet.

Exclusion Criteria:

* Individuals who have a reading disorder, cognitive impairment, dementia, or intellectual disabilities
* Individuals who are participating in any research studies
* Individuals who had participated in our previous feasibility study of the same intervention

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Brief Coping Orientation to Problems Experienced Inventory (Brief-COPE) | Immediately and two months after completion of the intervention in the experimental group
  Change in participants' coping strategies, as assessed using the Brief-COPE. This measure has 28 items and is a commonly used self-report measure of coping strategies. The Chinese version of the Brief-COPE had excellent internal consistency, test-retest reliability and content validity. Higher scores indicate more significant use of that specific coping strategy.

SECONDARY OUTCOMES:
Dissociative Experiences Scale-Taxon (DES-T) | Immediately and two months after completion of the intervention in the experimental group
  Change in participants' pathological dissociative experiences, as assessed using the DES-T. This measure has 8 items and can be used to screen for pathological dissociative experiences. The Chinese version of the DES-T demonstrated good construct validity and good discriminant validity between participants with and without clinically diagnosed dissociative disorders, with a cut-off score of 20. Higher scores indicate more frequent dissociative symptoms.

OTHER OUTCOMES:
Emotion Regulation Questionnaire (ERQ) | Immediately and two months after completion of the intervention in the experimental group
  Change in participants' emotion regulation, as assessed using the ERQ. This measure has 10 items and is a self-report measure of emotion regulation. It has good internal consistency and established construct validity. The Chinese version of the ERQ also demonstrates good internal consistency and construct validity. Higher scores indicate greater use of that particular emotion regulation strategy.
General Self-Efficacy Scale (GSES) | Immediately and two months after completion of the intervention in the experimental group
  Change in participants' self-efficacy, as assessed using the GSES. This measure has 10 items and is to assess respondents' level of self-efficacy by using a 4-point Likert scale to rate their self-beliefs to cope with adversities in different life situations. The total score ranges from 10 to 40, with the higher the score indicating the higher their perceived competence in managing difficult demands in life. The Chinese version of the GSES also demonstrated excellent internal consistency and good construct validity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam SKK, Fung HW. Can dissociative symptoms be explained by coping and emotion regulation? A longitudinal investigation. Psychol Trauma. 2025 Nov;17(8):1691-1698. doi: 10.1037/tra0001713. Epub 2024 Jun 20. PMID 38900513